CLINICAL TRIAL: NCT02010957
Title: ￼Combined 18F-Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) and Metomidate Imaging for Adrenal Neoplasia (FAMIAN-Study) - a Diagnostic Study
Brief Title: Combined FDG-PET and 123I-Iodometomidate Imaging for Adrenal Neoplasia
Acronym: FAMIAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stop of tracer production by company, unavailability of 123I Iodometomidate at most study centers, slow recruitment
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: German Research Foundation (Other); Steroid Metabolism Analysis Core, University of Birmingham (Unknown); EU FP7 ENSAT Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAMIAN (KS8-341); 2012-003604-13 (EudraCT Number)
Record Dates: First submitted 2013-12-04; First posted 2013-12-13 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Adrenal Neoplasia
Keywords: 123I Iodometomidate imaging; 18F FDG positron emission tomography; Adrenal tumour; Adrenal neoplasia
MeSH Terms: conditions — Adrenal Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FDG positron emission tomography and Iodometomidate imaging (Experimental): Combined FDG PET and Iodometomidate imaging prior adrenal surgery of uncertain adrenal neoplasms
  Interventions: Other: FDG positron emission tomography; Other: Iodometomidate imaging

INTERVENTIONS:
Other: FDG positron emission tomography — 2 consecutive imaging studies (diagnostic study) within 1-2 weeks: FDG-PET and 123I-Iodometomidate imaging in patients with an indeterminate adrenal neoplasm
  Other Names: FDG PET
Other: Iodometomidate imaging — 2 consecutive imaging studies (diagnostic study) within 1-2 weeks: FDG-PET and 123I-Iodometomidate imaging in patients with an indeterminate adrenal neoplasm
  Other Names: IMTO imaging; 123I-Iodometomidate imaging

SUMMARY:
Adrenal masses are highly prevalent and detected with high frequency by conventional imaging. Conventional imaging often fails to rule out a malignant lesion. Accordingly, most hormonally inactive adrenal masses removed by surgery are benign adenomas for which surgical removal is unnecessary and poses an avoidable risk to the patients. We hypothesize that the combination of FDG-PET and 123I-Iodometomidate imaging has the potential to noninvasively identify benign adrenocortical adenomas with high accuracy, thereby avoiding unnecessary surgery. Uptake of 123I-Iodometomidate by the adrenal mass demonstrates the presence of CYP 11B enzymes which specifically bind metomidate with high avidity establishing the adrenocortical origin of the lesion, while low uptake of FDG-PET in an adrenocortical lesion establishes its benign nature and excludes the presence of adrenocortical cancer (ACC). The proposed trial will assess the sensitivity, specificity, positive and negative predictive value of the combined imaging for the diagnosis of adrenocortical adenoma. A secondary focus is on the performance of the combined test for differentiating ACC from non-ACC lesions. We expect that the results of our trial will help to greatly reduce the need for surgery in hormonally inactive adrenal masses.

DETAILED DESCRIPTION:
Histopathology of a surgically removed adrenal mass by an expert surgeon is considered to be the gold standard for the differential diagnosis of an adrenal neoplasia. Thus we will only recruit patients scheduled for surgery for an adrenal mass of uncertain origin. Patients will be eligible for the trial when an adrenal mass has been discovered and standard imaging (CT and/or MRI) has not led to a clear characterization of the malignant potential of the lesion (Hounsfield units in unenhanced CT ≥10). In addition, patients with adrenal neoplasia will be only recruited when a hormonally active lesion has been excluded and surgery is planned because of a perceived risk of malignancy. Patients will be evaluated by both [123I]Iodometomidate SPECT/CT and [18F]fluorodeoxyglucose PET/CT. Computed tomography will be performed as low dose CT of the adrenal region. Imaging can be started with either [123I]Iodometomidate SPECT/CT or [18F]fluoro- deoxyglucose PET/CT and can be performed at two consecutive days. The time interval between [123I]Iodometomidate SPECT/CT and [18F]fluorodeoxyglucose PET/CT should not exceed 6 weeks. Patients will have a follow up visit 2-4 weeks after [123I]Iodometomidate SPECT/CT and [18F]fluorodeoxyglucose PET/CT (or immediately before surgery, if earlier than 2 weeks post imaging). Thirty days after surgery patients will be contacted by phone for assessment of adverse events related to surgery.

ELIGIBILITY:
Inclusion Criteria

* Patients aged >= 30 years
* with a solid indeterminate adrenal mass with a diameter > 3 cm or an increase in tumor diameter of > 1 cm after the initial evaluation
* with an attenuation value of the adrenal tumor >= 10 Hounsfield units (HU) in unenhanced computerized tomography (CT)
* scheduled for surgery or biopsy within 3 months
* Written informed consent
* ECOG performance status 0-2
* Effective contraception in female patients of childbearing potential
* Negative pregnancy test in women of childbearing potiential
* Ability to comply with protocol procedures

Exclusion Criteria

* Pregnancy or breast feeding
* Patient unfit or unwilling to undergo surgery / biopsy
* Diagnosis of pheochromocytoma
* Diagnosis of primary hyperaldosteronism
* Diagnosis of Cushing´s syndrome

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Specificity of combined FDG-PET and 123I-IMTO imaging for diagnosing adrenocortical adenoma | within 1 to 2 weeks (minimum 2 days, maximum 6 weeks)
  Diagnostic study with combined FDG-PET and 123I-IMTO imaging in which an indeterminate adrenal mass with negative FDG-PET test (FDG-) and positive 123I-IMTO test (IMTO+) is diagnosed as a benign adrenocortical adenoma (AA+). Primary efficacy endpoint: Specificity (rate estimation) of the diagnostic AA test and likelihood ratio of a positive diagnostic test (using rate estimation of the sensitivity). The outcome measure does not assess a change but the diagnostic accuracy of both FDG-PET and IMTO imaging.

SECONDARY OUTCOMES:
Sensitivity of combined FDG-PET and 123I-IMTO imaging for diagnosing adrenocortical adenoma | within 1 to 2 weeks (minimum 2 days, maximum 6 weeks)
  Sensitivity of the diagnostic adrenocortical adenoma (AA) test and likelihood ratio of a negative diagnostic AA test, a priori rates of AA, adrenocortical cancer (ACC) and other benign as well as malignant indeterminate adrenal neoplasias. Detection rates similar to sensitivity and specificity for ACC and indeterminate adrenal neoplasias other than AA and ACC of combined 18F-FDG-PET imaging and 123I-Iodometomidate imaging in identifying ACC. Predictive values will be determined and economic analysis of cost effectiveness of diagnostic evaluation versus surgery for all indeterminate lesions will be performed. The outcome measure does not assess a change but the diagnostic accuracy of both FDG-PET and IMTO imaging.

OTHER OUTCOMES:
Assessment of safety of 123I-IMTO imaging | 2 to 4 weeks after IMTO imaging
  Adverse events as well as standard routine parameter changes from before imaging to prior surgery will be assessed (plus follow up analysis until 30 days after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Hahner, Prof. Dr., Principal Investigator — University of Wuerzburg
Locations (6):
- Germany (6):
  - Charité Universiaetsmedizin, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinik Leipzig, Leipzig
  - Universitaetsmedizin Mainz, Mainz
  - Klinikum der Universitaet Muenchen, München
  - University Hospital Wuerzburg, Würzburg

REFERENCES:
- [Background] Hahner S, Kreissl MC, Fassnacht M, Haenscheid H, Bock S, Verburg FA, Knoedler P, Lang K, Reiners C, Buck AK, Allolio B, Schirbel A. Functional characterization of adrenal lesions using [123I]IMTO-SPECT/CT. J Clin Endocrinol Metab. 2013 Apr;98(4):1508-18. doi: 10.1210/jc.2012-3045. Epub 2013 Feb 20. PMID 23426614
- [Background] Hahner S, Stuermer A, Kreissl M, Reiners C, Fassnacht M, Haenscheid H, Beuschlein F, Zink M, Lang K, Allolio B, Schirbel A. [123 I]Iodometomidate for molecular imaging of adrenocortical cytochrome P450 family 11B enzymes. J Clin Endocrinol Metab. 2008 Jun;93(6):2358-65. doi: 10.1210/jc.2008-0050. Epub 2008 Apr 8. PMID 18397978
- [Result] https://doi.org/10.1016/j.ebiom.2025.105735
- [Derived] Hahner S, Hartrampf P, Beuschlein F, Miederer M, Miehle K, Schlotelburg W, Fuss CT, Pfluger T, Fottner C, Tonjes A, Herrmann K, Amthauer H, Reincke M, Schreckenberger M, Sabri O, Werner J, Reuter M, Kircher S, Arlt W, Fassnacht M, Konrad Buck A, Muller HH, Schirbel A; FAMIAN investigators. Combined [18F]Fluorodeoxyglucose PET and [123I]Iodometomidate-SPECT for diagnostic evaluation of indeterminate adrenal neoplasias-the cross-sectional diagnostic test accuracy study FAMIAN. EBioMedicine. 2025 Jun;116:105735. doi: 10.1016/j.ebiom.2025.105735. Epub 2025 May 20. PMID 40398350